CLINICAL TRIAL: NCT05021081
Title: Visual Performance of Senofilcon A With and Without a New UV/HEV-filter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6463
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Visual Performance

STUDY DESIGN:
Intervention Model Description: In Phase 2, subjects will be randomized to a contralateral sequence where the study lenses will be worn throughout the duration of the study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): For Phase 2, eligible subjects that are enrolled will be randomized to the Test/Control contralateral sequence.
  Interventions: Device: TRP-200; Device: ACUVUE Oasys 1-Day
- CONTROL/TEST (Experimental): For Phase 2, eligible subjects that are enrolled will be randomized to the Control/Test contralateral sequence.
  Interventions: Device: TRP-200; Device: ACUVUE Oasys 1-Day

INTERVENTIONS:
Device: TRP-200 — JJVC Investigational Contact Lens
  Other Names: TEST
Device: ACUVUE Oasys 1-Day — JJVC Marketed Contact Lens
  Other Names: CONTROL

SUMMARY:
This study will occur in two non-dispensing phases: Phase 1 is a non-randomized, non-masked, non-dispensing study where subjects will wear their own contact lenses for approximately 1 hour. Phase 2 is a controlled, randomized, double-masked, contralateral non-dispensing study where the study lenses will be worn in a daily wear modality for approximately 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. For Phase I be between 18-39 (inclusive) years of age at the time of screening.
  4. For Phase II be between 18 and 70 (inclusive) years of age at the time of screening.
  5. By self-report, habitually wear spherical silicone hydrogel soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.
  6. Possess a wearable pair of spectacles that provide correction for distance vision.
  7. Habitual spherical contact lens powers must be between -1.00 D and -6.00 D (inclusive) in each eye.
  8. For Phase I, habitual contact lenses must provide at least 20/20 acuity OD and OS.
  9. For Phase II, the spherical equivalent of the subject's vertex-corrected distance refraction must be between -1.00 D and -6.00 D (inclusive) in each eye.
  10. For Phase II, the magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be between 0.00 D and 1.00 D (inclusive) in each eye.
  11. For Phase II, the best corrected, monocular, distance visual acuity must be 20/25 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or lactating.
  2. Be currently using any ocular medications or have any ocular infection of any type.
  3. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures.
  4. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
  5. Be currently wearing monovision or multifocal contact lenses.
  6. Be currently wearing lenses in an extended wear modality.
  7. Have participated in a contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  8. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
  9. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
  10. Have a history of strabismus or amblyopia.
  11. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
  12. Have had any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).
  13. Have signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar).
  14. Have a history of eyelid injury, surgery or procedure that resulted in abnormal eyelid position or movement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Phase I, 20 subjects were enrolled and completed this Phase. In Phase 2, 62 subjects were enrolled. Of those enrolled in Phase 2, all 62 were dispensed at least 1 study lens. Of those dispensed, 60 subjects completed Phase 2 while 2 subjects were discontinued from Phase 2.
  Phase I and Phase II are mutually exclusive. Data collected from Phase I was used to validate the glare light source for evaluating the primary and secondary endpoints in Phase II.
Units Other Than Participants: Eyes
Groups:
- OD: Test (Senofilcon A C3) /OS: Control (Senofilcon A C3) (Phase 2): Subjects randomized to this sequence received the Test lens on the right eye and received the Control lens on the left eye
- OD: Control (Senofilcon A C3) / OS: Test (Senofilcon A C3) (Phase 2): Subjects randomized to this sequence received the Control lens on the right eye and received the Test lens on the left eye
- Subjects' Own Contact Lens (Phase 1): Subjects enrolled into this phase used the following marketed contact lenses: senofilcon A (1-Day), senofilcon A (2-week reusable), senofilcon A C3, lotrafilcon B, comifilcon A, somofilcon A, delefilcon A, and stenfilcon A
Period: Phase 1
Arm/Group | OD: Test (Senofilcon A C3) /OS: Control (Senofilcon A C3) (Phase 2) | OD: Control (Senofilcon A C3) / OS: Test (Senofilcon A C3) (Phase 2) | Subjects' Own Contact Lens (Phase 1)
Started | 0; 0 Eyes | 0; 0 Eyes | 20; 40 Eyes
Completed | 0; 0 Eyes | 0; 0 Eyes | 20; 40 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes
Period: Phase 2
Arm/Group | OD: Test (Senofilcon A C3) /OS: Control (Senofilcon A C3) (Phase 2) | OD: Control (Senofilcon A C3) / OS: Test (Senofilcon A C3) (Phase 2) | Subjects' Own Contact Lens (Phase 1)
Started | 31; 62 Eyes | 31; 62 Eyes | 0; 0 Eyes
Completed | 30; 60 Eyes | 30; 60 Eyes | 0; 0 Eyes
Not Completed | 1; 2 Eyes | 1; 2 Eyes | 0; 0 Eyes
Not completed — Subject enrolled in error | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled and completed in Phase 1. All subjects dispensed in Phase 2.
Groups:
- Phase 1: Phase 1 was a non-randomized design where subjects wore their own contact lenses
- Phase 2: Phase 2 was a randomized design with two test articles
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 20 | 62 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (5.62) | 38.6 (14.07) | 35.2 (13.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 50 | 66
  Male | 4 | 12 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 4 | 5
  Black or African American | 2 | 7 | 9
  White | 16 | 51 | 67
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 62 | 82

OUTCOME MEASURES:

1. Primary Outcome: Photopic Contrast Sensitivity at 6 Cpd
Description: Photopic (~120 cd/m2) contrast sensitivity at 6 cpd was measured on the right eye only with and without a broadband glare source (with glare followed after without glare). Testing included 8 reversals with the last 4 being averaged to provide the contrast threshold. If the reduction (indicating worse contrast sensitivity) in the estimated mean due to the glare source was about 0.1 log units, then it can be concluded that the glare light source was effective and the study can move to Phase 2.
Time Frame: Post screening up to 1 hour during Phase 1
Population: All subjects that completed Phase 1 without a major protocol deviation excluding subjects recording an increase in photopic contrast sensitivity with the glare source.
Measure: Mean (Standard Deviation); unit: Log Unit
Units Other Than Participants: Eyes
Groups:
- With Glare: Subjects with photopic contrast sensitivity measured with a broadband glare source during Phase 1.
- Without Glare: Subject with photopic contrast sensitivity measured without a broadband glare source during Phase 1.
Arm/Group | With Glare | Without Glare
Number analyzed (Participants) | 15 | 15
Number analyzed (Eyes) | 15 | 15
Log Unit | 1.46 (0.317) | 1.91 (0.373)
Statistical Analysis 1: Comparison: With Glare vs Without Glare; The sample size was chosen based on resources in conjunction, subject matter experts, and any available literature. To help ensure the glare source intensity, a small pilot investigation per the ANSI Z80.12-2007 standard was interpreted to be about 20 subjects to complete Phase 1, which should be sufficient to evaluate the mean photopic contrast sensitivity with and without the glare source; Test type: Other — The least-square means (i.e., adjusted means) of photopic contrast sensitivity at 6 cpd was estimated separately under conditions with glare source and without glare source. This endpoint was not statistically tested, and consequentially statistical interferences was not made; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = -0.45, 95% CI 2-sided [-0.70 to -0.21], Standard Error of Mean 0.114 — Least-square Mean difference was calculated as With glare minus Without glare

2. Primary Outcome: Mesopic Contrast Sensitivity at 6 Cpd
Description: Mesopic (~3 cd/m2) contrast sensitivity at 6 cpd was measured on the right eye only with and without a broadband glare source (with glare followed after without glare). Testing included 8 reversals with the last 4 being averaged to provide the contrast threshold. If the reduction (indicating worse contrast sensitivity) in the estimated mean due to the glare source was about 0.1 log units, then it can be concluded that the glare light source was effective and the study can move to Phase 2.
Time Frame: Post screening up to 1 hour during Phase 1
Population: All subjects completed Phase 1 without a major protocol deviation excluding subjects recording an increase in mesopic contrast sensitivity with the glare source.
Measure: Mean (Standard Deviation); unit: Log Unit
Units Other Than Participants: Eyes
Arm/Group | With Glare | Without Glare
Number analyzed (Participants) | 14 | 14
Number analyzed (Eyes) | 14 | 14
Log Unit | 0.70 (0.328) | 1.29 (0.498)
Statistical Analysis 1: Comparison: With Glare vs Without Glare; The sample size was chosen based on resources in conjunction, subject matter experts, and any available literature. To help ensure the glare source intensity, a small pilot investigation per the ANSI Z80.12-2007 standard was interpreted to be about 20 subjects to complete Phase 1, which should be sufficient to evaluate the mean mesopic contrast sensitivity with and without the glare source; Test type: Other — The least-square means (i.e., adjusted means) of mesopic contrast sensitivity at 6 cpd was estimated separately under conditions with glare source and without glare source. This endpoint was not statistically tested, and consequentially statistical interferences was not made; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = -0.58, 95% CI 2-sided [-0.81 to -0.36], Standard Error of Mean 0.102 — Least-square Mean difference was calculated as With glare minus Without glare

3. Primary Outcome: Photopic Resolution Acuity Using Landolt C's With a Glare Source
Description: Photopic resolution acuity using Landolt C's was measured separately for the right (OD) and left (OS) eyes, using an arcminute scale under bright light conditions (~120 cd/m2) with a broadband glare source. The photopic resolution acuity on arcminute scale was converted to logMAR scale for the analysis purpose using a log transformation. Lower values indicate better acuity.
Time Frame: At least 5 minutes post lens fitting up to 2 hours during Phase 2
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Test (Senofilcon A C3): Subject eyes that wore the Test lens during the study.
- Control (Senofilcon A C3): Subject eyes that wore the Control lens during the study.
Arm/Group | Test (Senofilcon A C3) | Control (Senofilcon A C3)
Number analyzed (Participants) | 62 | 62
Number analyzed (Eyes) | 62 | 62
logMAR | 0.01 (0.191) | -0.01 (0.158)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3) vs Control (Senofilcon A C3); Given no historical data is available, the sample size was not determined based on any empirical sample size calculation. A power analysis was conducted using a paired sample t-test (exact method) with a 2-sided type I error rate 0.05 to estimate statistical power based on different assumptions. The power analysis showed that the statistical power for testing superiority would be approximately 80% or higher with the effect size of -0.05 (mean difference: Test minus Control); Test type: Superiority — Superiority was declared if the upper bound of the 2-sided 95% confidence interval of the mean difference was below 0; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = 0.019, 95% CI 2-sided [-0.029 to 0.068], Standard Error of Mean 0.024 — Least-square Mean difference was calculated as Test minus Control

4. Secondary Outcome: Photopic Contrast Sensitivity With a Glare Source
Description: Photopic contrast sensitivity was measured for the right (OD) and left (OS) eyes separately under bright light conditions (~120 cd/m2) with a broadband glare source. Testing included 8 reversals with the last 4 being averaged to provide the contrast threshold. The area under the log contrast sensitivity function (AULCSF) was derived for the analysis using the trapezoidal rule. Higher AULCSF values indicate better contrast sensitivity.
Time Frame: At least 5 minutes post lens fitting up to 2 hours during Phase 2
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A C3) | Control (Senofilcon A C3)
Number analyzed (Participants) | 62 | 62
Number analyzed (Eyes) | 62 | 62
Units on a scale | 1.18 (0.248) | 1.21 (0.250)

5. Secondary Outcome: Mesopic Contrast Sensitivity With a Glare Source
Description: Mesopic contrast sensitivity was measured for the right (OD) and left (OS) eyes separately under dim light conditions (less than or equal 3 cd/m2) with a broadband glare source. Testing included 8 reversals with the last 4 being averaged to provide the contrast threshold. The area under the log contrast sensitivity function (AULCSF) was derived for the analysis using the trapezoidal rule. Higher AULCSF values indicate better contrast sensitivity.
Time Frame: At least 5 minutes post lens fitting up to 2 hours during Phase 2
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A C3) | Control (Senofilcon A C3)
Number analyzed (Participants) | 62 | 62
Number analyzed (Eyes) | 62 | 62
Units on a scale | 0.71 (0.212) | 0.72 (0.232)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; Phase 1 was approximately 1 hour per subject. Phase 2 was approximately 3 hours per subject.
Groups:
- Phase 1 - Senofilcon A (1-Day): Subjects enrolled into Phase I of the study with senofilcon A (1-Day) as their own contact lens.
- Phase 1 - Senofilcon A (2-week Reusable): Subjects enrolled into Phase I of the study with senofilcon A (2-week reusable) as their own contact lens.
- Phase 1 - Senofilcon A C3: Subjects enrolled into Phase I of the study with senofilcon A C3 as their own contact lens.
- Phase 1 - Lotrafilcon B: Subjects enrolled into Phase I of the study with lotrafilcon B as their own contact lens.
- Phase 1 - Comifilcon A: Subjects enrolled into Phase I of the study with comifilcon A as their own contact lens.
- Phase 1 - Somofilcon A: Subjects enrolled into Phase I of the study with somofilcon A as their own contact lens.
- Phase 1 -Delefilcon A: Subjects enrolled into Phase I of the study with delefilcon A as their own contact lens.
- Phase 1 -Stenfilcon A: Subjects enrolled into Phase I of the study with stenfilcon A as their own contact lens.
- Phase 2 - Control (Senofilcon A C3): Subjects that wore the Control lens in either eye during Phase 2 of the study.
- Phase 2 - Test (Senofilcon A C3): Subjects that wore the Test lens in either eye during Phase 2 of the study.
Arm/Group | Phase 1 - Senofilcon A (1-Day) | Phase 1 - Senofilcon A (2-week Reusable) | Phase 1 - Senofilcon A C3 | Phase 1 - Lotrafilcon B | Phase 1 - Comifilcon A | Phase 1 - Somofilcon A | Phase 1 -Delefilcon A | Phase 1 -Stenfilcon A | Phase 2 - Control (Senofilcon A C3) | Phase 2 - Test (Senofilcon A C3)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/2 | 0/1 | 0/1 | 0/4 | 0/2 | 0/3 | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/2 | 0/1 | 0/1 | 0/4 | 0/2 | 0/3 | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/2 | 0/1 | 0/1 | 0/4 | 0/2 | 0/3 | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT05021081/Prot_SAP_000.pdf